CLINICAL TRIAL: NCT03600974
Title: A New System for Diagnosis and Treatment of Gastroesophageal Refulx Diseases : Based on Endoscopy, pH Parameter, Impedence Parameter, High Resolution Manometry and Psychology
Brief Title: A New System for GERD Diagnosis and Treatment
Acronym: EAISMLP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Guo Zihao, Principal Investigator, Capital Medical University
Other Study IDs: xhnk002
Record Dates: First submitted 2018-06-21; First posted 2018-07-26 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Omeprazole; Lansoprazole; Rabeprazole; Esomeprazole; Pantoprazole; mosapride; Domperidone; Neurotransmitter Agents; flupentixol, melitracen drug combination; Citalopram

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (14):
- Endoscopy-E(+): Subjects with positive endoscopy finding:erosive esophagitis or Barrett esophagus.For subjects of this group, PPIs, Stretta,Laparoscopic Nissen fundoplication is considered.
  Interventions: Procedure: Stretta; Procedure: Laparoscopic Nissen fundoplication; Drug: PPI
- Endoscopy-E(-): Subjects with negative endoscopy finding:NERD.
- Acid-A(+): Subjects with DeMeester scores>14.72.For subjects of this group, PPIs, Stretta,Laparoscopic Nissen fundoplication is considered.
  Interventions: Procedure: Stretta; Procedure: Laparoscopic Nissen fundoplication; Drug: PPI
- Acid-A(-): Subjects with DeMeester scores<14.72
- impedance-I（+）W/S: Subjects with total reflux number > 80 in 24h pH-impedance monitoring. W means weakly acid reflux account for above 50% in total reflux number. G means gas reflux account for above 50% in total reflux number.For subjects of this group,probiotic agent is considered.
  Interventions: Drug: Probiotic Agent
- impedance-I（-）: Subjects with total reflux number < 80 in 24h pH-impedance monitoring.
- Reflux-symptom association-S(+): Subjects with positive reflux-symptom association.For subjects of this group, PPIs, Stretta, neuromodulators are considered.
  Interventions: Procedure: Stretta; Drug: PPI; Drug: Neuromodulators
- Reflux-symptom association-S(-): Subjects with negative reflux-symptom association
- motility-M(+): Subjects with motility disorders according to Chicago v3.0.For subjects of this group, prokinetic motility agents are considered.
  Interventions: Drug: Prokinetic Motility Agents
- motility-M(-): Subjects without motility disorders according to Chicago v3.0
- lower oesophageal sphincter-L(+): Subjects with abnormal LES pressure or EGJ type III or hiatus hernia.For subjects of this group, Stretta,Laparoscopic Nissen fundoplication is considered.
  Interventions: Procedure: Stretta; Procedure: Laparoscopic Nissen fundoplication
- lower oesophageal sphincter-L(-): Subjects with normal LES pressure and EGJ type I~II
- psychology-P(+): Subjects with normal psychology condition.For subjects of this group,neuromodulators are considered.
  Interventions: Drug: Neuromodulators
- psychology-P(-): Subjects with abnormal psychology condition

INTERVENTIONS:
Procedure: Stretta — Stretta for Endoscopy-E(+),Acid-A(+),Reflux-symptom association-S(+) or lower oesophageal sphincter-L(+) group
  Groups: Acid-A(+); Endoscopy-E(+); Reflux-symptom association-S(+); lower oesophageal sphincter-L(+)
Procedure: Laparoscopic Nissen fundoplication — Laparoscopic Nissen fundoplication for E(+),A(+) or L(+) group
  Groups: Acid-A(+); Endoscopy-E(+); lower oesophageal sphincter-L(+)
Drug: Probiotic Agent — Probiotic Agent for I(+)G/W；Live Bacillus Licheniformis Cranules 0.5g bid； Bifidbacterium 0.63g bid
  Other Names: Live Bacillus Licheniformis Cranules; Bifidbacterium
  Groups: impedance-I（+）W/S
Drug: PPI — PPIs for A(+),E(+)or S(+) patients: Nexium 20mg Qd/Bid;Lansoprazole 30mg Qd/Bid；omeprazole 10mg-30mg Qd-Bid;Rabeprazole 10mg Qd/Bid;Esomeprazole 20mg Qd/Bid;Pantoprazole 40mg Qd/Bid
  Other Names: omeprazole; lansoprazole; Rabeprazole; Esomeprazole; Pantoprazole
  Groups: Acid-A(+); Endoscopy-E(+); Reflux-symptom association-S(+)
Drug: Prokinetic Motility Agents — Prokinetic Motility Agents for M(+) group; Mosapride 5mg Tid; Domperidone 10mg Tid
  Other Names: Mosapride; Domperidone
  Groups: motility-M(+)
Drug: Neuromodulators — Neuromodulators for P(+) or S(+);Flupentixol and Melitracen 1# bid;
  Other Names: Flupentixol and Melitracen; Citalopram
  Groups: Reflux-symptom association-S(+); psychology-P(+)

SUMMARY:
This is a pilot study measuring a new diagnosis and treatment system "EAISMLP" in adult patients with gastroesophageal reflux disease (GERD).

DETAILED DESCRIPTION:
The investigators created a new diagnosis and treatment system for gastroesophageal reflux disease (GERD). The system based on endoscopy, 24h esophageal pH-impedance monitoring, esophagus high resolution manometry and psycological condition.the investigators named it as "EAISMLP" symptom. Each letter in "EAISMLP" is responsible for a typical character and treatment. Subjects will be subtyped according to "EAISMLP" system and underwent treatment, and will be follow up for 6 months and 1 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female aged ≥18 years
2. Subjects with refractory reflux symptoms to PPIs standard treatment as follows:

   2.1 Ongoing heartburn symptom with or without these GERD-related symptoms : Regurgitation, Non-cardiac chest pain, Epigastric pain, Belching, Bloating, Satiety, Sore throat, Cough, Laryngitis, Hoarseness, Nausea, Vomiting, Dysphagia, Odynophagia, Weight loss.

   2.2 Ongoing heartburn symptom with or without erosion ≥ grade A according to LA Classification.
3. Decided to participate and signed on an informed consent form willingly.

Exclusion Criteria:

1. Existence of upper gastrointestinal bleeding or active gastroduodenal ulcer at screening.
2. History of operation in esophagus, stomach or duodenum.
3. Primary esophageal motility disease, Achalasia, Scleroderma, Esophageal/ pyloric stricture, Primary esophageal spasm, Barrett's esophagus ≥ 3 cm, Zollinger-Ellison syndrome.
4. Infectious or inflammatory bowel disease, Severe malabsorption, Severe chronic heart failure, cardiovascular disease, renal failure, COPD, asthma, liver cirrhosis.
5. History of cancer within 5 years, except completely recovered skin cancer ALT or AST ≥ Upper limit of normal range X 3.
6. Need antibiotics due to severe infection.
7. Pregnant or breast-feeding women.
8. Conversation impairment because of alcohol, drug addiction or mental illness, etc.
9. Inability to record diary card
10. In investigator's judgement

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with refractory gastroesophageal refulx symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Satisfaction of the "EAISMLP system" on GERD symptoms assessed by the HRQL scores. | Change from Baseline HRQL scores at 1 month;Change from Baseline HRQL scores at 2 months;Change from Baseline HRQL scores at 6 months;Change from Baseline HRQL scores at 1 year
  mean improvement in the GERD-health-related quality of life (HRQL) scores. Scale ranges 0-50 points, the lower score means the better efficacy.

SECONDARY OUTCOMES:
Satisfaction of the "EAISMLP system" on life quality assessed by the SF-36 scores. | Change from Baseline SF-36 scores at 1 month;Change from Baseline SF-36 scores at 2 months;Change from Baseline SF-36 scores at 6 months;Change from Baseline SF-36 scores at 1 year
  mean improvement in SF-36 scores.Scale ranges 0-100 points, the higher score means the better efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Chuan Zhang, MD, Study Chair — Gatroenterology department,Beijing Tong Ren Hospital, Capital Medical University

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be avialable within 1 months of study completion.
Access Criteria: Data access requests will be reviewed by an external independant Review Panel. Requestors will be required to sign a Data Access Agreement.